CLINICAL TRIAL: NCT05734196
Title: The ENERGY Study: An Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INZ-701 in Infants With Ectonucleotide Pyrophosphatase/ Phosphodiesterase 1 (ENPP1) Deficiency or ATP-binding Cassette Sub-family C Member 6 (ABCC6) Deficiency
Brief Title: The ENERGY Study: Evaluation of Safety and Tolerability of INZ-701 in Infants With ENPP1 Deficiency or ABCC6 Deficiency
Acronym: ENERGY
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inozyme Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INZ701-104
Record Dates: First submitted 2023-01-26; First posted 2023-02-17 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Ectonucleotide Pyrophosphatase/phosphodiesterase1 Deficiency; Autosomal Recessive Hypophosphatemic Rickets; Generalized Arterial Calcification of Infancy; ATP-Binding Cassette Subfamily C Member 6 Deficiency; Pseudoxanthoma Elasticum
Keywords: ectonucleotide pyrophosphatase/phosphodiesterase1 deficiency; hypopyrophosphatemia; ENPP1; Generalized Arterial Calcification of Infancy; GACI; Autosomal Recessive Hypophosphatemic Rickets Type 2; ARHR2; ATP-Binding Cassette Subfamily C Member 6 Deficiency; ABCC6; Pseudoxanthoma elasticum; PXE
MeSH Terms: conditions — Hypophosphatemic Rickets, Autosomal Recessive, 1; Arterial calcification of infancy; Pseudoxanthoma Elasticum

STUDY DESIGN:
Intervention Model Description: Study INZ701-104 is a Phase 1b, open-label study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of INZ-701 in infant study participants with ENPP1 Deficiency or with ABCC6 Deficiency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INZ-701 (Experimental): The first 2 study participants will receive 1 dose of 0.2 mg/kg on Day 1 and start at Dose Level A (0.2 mg/kg twice weekly) on Day 8.
  The Data Review Committee (DRC) comprised of representatives of the Sponsor, the study Investigators, and a physician who is a subject matter expert not affiliated with the study or Sponsor, will review the safety data of the first study participant through Day 8. Contingent upon this review, the Sponsor will decide if additional study participants can begin receiving INZ-701.
  After the second study participant completes Day 32, the DRC will perform a cumulative review of safety and PK/PD data and will make dosing recommendations, for example, modifying the dose of the ongoing study participants and/or changing the starting dose for future participants.
  Dose Level A: 0.2 mg/kg twice weekly
  Dose Level B: 0.6 mg/kg twice weekly
  Dose Level C: 0.2 mg/kg once weekly
  Dose Level D: 0.6 mg/kg once weekly
  Dose Level E: 1.8 mg/kg once weekly
  Interventions: Drug: INZ-701

INTERVENTIONS:
Drug: INZ-701 — Recombinant fusion protein that contains the extracellular domains of human ENPP1 coupled with an Fc fragment from an immunoglobulin gamma-1 (IgG1) antibody.
  Other Names: (rhENPP1-Fc).

SUMMARY:
The primary purpose of Study INZ701-104 (the ENERGY study) is to assess the safety and tolerability of INZ-701 in infants with ENPP1 Deficiency or with ABCC6 Deficiency.

DETAILED DESCRIPTION:
INZ-701 is an ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) enzyme replacement therapy in development for the treatment of the ultra-rare genetic disorder, ENPP1 Deficiency or with ABCC6 Deficiency.

Study INZ701-104 (the ENERGY study) is a Phase 1b, open-label study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of INZ-701 in infant study participants with ENPP1 Deficiency or ABCC6 Deficiency.

The study will consist of up to a 60-day Screening Period, a 52-week Treatment Period during which study participants will receive INZ-701, an Extension Period during which participants may continue to receive INZ-701 until it is commercially available in the country where the participant resides, or until an alternative study of INZ-701 is available, and an End of Treatment (EOT) visit 30 days after the last dose of INZ-701. Upon treatment discontinuation, participants will continue to be followed for their ongoing disposition for survival outcome at least quarterly through the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Caregiver(s) must provide written or electronic consent after the nature of the study has been explained, and prior to any research-related procedures, per International Council for Harmonisation (ICH) Good Clinical Practice (GCP)
2. Study participant must have a confirmed post-natal molecular genetic diagnosis of ENPP1 Deficiency or ABCC6 Deficiency with biallelic mutations (ie, homozygous or compound heterozygous) performed by a College of American Pathologists/Clinical Laboratory Improvement Amendments (CAP/CLIA) certified laboratory
3. Study participants must have clinical manifestations of GACI or GACI-2, which may include, but are not limited to, pathologic ectopic calcification, heart failure, respiratory distress, edema, cyanosis, hypertension, and cardiomegaly
4. Study participant must be male or female from birth to <1 year of age at Baseline (Day 1)
5. Study participant must weigh ≥0.5 kg at the time of the first dose of INZ-701 in this study
6. In the opinion of the Investigator, the study participant must be able to complete all aspects of the study
7. Study participant's caregiver(s) must agree to provide access to their child's relevant medical records

Exclusion Criteria:

1. In the opinion of the Investigator, presence of any clinically significant disease or laboratory abnormality (outside of those considered associated with the diagnosis of ENPP1 Deficiency or ABCC6 Deficiency) that precludes study participation or may confound interpretation of study results, including known uncontrolled thyroid disease or unrelated connective tissue, bone, mineral, or muscle disease
2. Care has been withdrawn or study participant is receiving end of life care or hospice only
3. Known malignancy
4. Known intolerance to INZ-701 or any of its excipients
5. Concurrent participation in another non-Inozyme interventional study
6. Receipt of any non-Inozyme investigational new drug within 5 half-lives of the last dose of the other investigational product or within 4 weeks prior to the first dose of INZ-701, whichever is longer, or use of an investigational device, through completion of participation in the study

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) | 52 weeks (Treatment Period)
  Treatment-emergent AEs are defined as any AE occurring from the first dose of INZ-701 through 30 days after the last dose of INZ-701.
Incidence of Anti-Drug Antibodies (ADA) | 52 weeks (Treatment Period)
  For each participant, the presence of ADAs will be assessed and, if present, further evaluation will determine specificity and subtypes.
Left Ventricular Ejection Fraction | 52 weeks (Treatment Period)
  For each participant, an echocardiogram will be collected, and used to assess heart function. (Including measurement of left ventricular ejection fraction), and to identify any other abnormalities, for example, calcification of heart valves.

SECONDARY OUTCOMES:
Change from Baseline in Plasma Inorganic Pyrophosphate (PPi) Levels | 52 weeks (Treatment Period)
  For each participant, plasma PPi will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.
Area under the Plasma Concentration versus Time Curve (AUC) of INZ-701 | 52 weeks (Treatment Period)
  For each participant, variation of concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.
Maximum Plasma Concentration (Cmax) of INZ-701 | 52 weeks (Treatment Period)
  For each participant, the maximum concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.
ENPP1 Activity | 52 weeks (Treatment Period)
  For each participant, the activity of INZ-701 in the serum will be measured via a series of blood samples obtained throughout the study, comparing the participant's baseline value over time.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Lai, MD, Study Director — Inozyme Pharma
Locations (7):
- United States (5):
  - Rady Children's Hospital, San Diego, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Utah, Salt Lake City, Utah
- Hospital Sant Joan de Déu, Barcelona, Spain
- Royal Manchester Children's Hospital, Manchester, United Kingdom